CLINICAL TRIAL: NCT00587106
Title: Studies of Neurological Paraneoplastic Syndromes
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Jerome Posner, MD, Memorial Sloan-Kettering Cancer Center
Other Study IDs: 88-044
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2009-03-30 (Estimated); Status verified 2009-03

CONDITIONS: Paraneoplastic Neurologic Degenerations (PNDs)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood and/or spinal fluid

GROUPS / COHORTS (1):
- 1: One cohort group of patient with PNDS or suspected PNDS

SUMMARY:
This study is for patients with cancer, a known paraneoplastic syndrome, or neurological problems that suggest a paraneoplastic syndrome.

DETAILED DESCRIPTION:
Patients usually go to their doctors with neurological complaints and later find they have cancer, a known paraneoplastic syndrome, or neurological problems that suggest a paraneoplastic syndrome. Paraneoplastic syndromes are rare conditions in which the immune system is involved in causing brain damage and fighting cancer.

Such patients with paraneoplastic neurologic degenerations(PNDs) may have autoantibodies, an antibody or protein the immune system creates that is directed against his or her own proteins. This study aims to better understand PNDS by:

* analyzing for autoantibodies in serum and cerebral spinal fluid
* analyzing for antigen specificity and for antigens in cancer tissue
* comparing PND autoantibodies with those in cancer patients but no PND
* comparing PND autoantibodies with those in PND patients but no cancer
* studying the immune performance of patients with PNDs

As this study is not a treatment study, tissues for this study will only come from procedures necessary for the patient's treatment.

ELIGIBILITY:
Inclusion Criteria:

* All adults are potentially eligible.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are selected from severals clinics within Memorial Sloan-Kettering Cancer Cetner
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 1988-04; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Increase understanding of PNDS | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Jerome Posner, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org